CLINICAL TRIAL: NCT06851104
Title: A Prospective Study of Cadonilimab in Hepatocellular Carcinoma After Radical Surgery With High Risk of Recurrence
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Professor, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PREVENT-3
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: hepatocellular carcinoma; hepatectomy; adjuvant; cadonilimab
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Patients with hepatocellular carcinoma after curative hepatectomy would be suggested to receive cadonilimab 10 mg/kg intravenous infusion (dissolved in 0.9% NaCl 250 mL, within 60 minutes) Q3W, until disease progression, death, intolerance to toxicity, withdrawal of informed consent, initiation of new anti-tumor treatment, or termination of treatment for other reasons specified in the protocol. The maximum treatment duration for cadonilimab is 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Patients with hepatocellular carcinoma after curative hepatectomy would receive cadonilimab 10 mg/kg intravenous infusion (dissolved in 0.9% NaCl 250 mL, within 60 minutes) Q3W, until disease progression, death, intolerance to toxicity, withdrawal of informed consent, initiation of new anti-tumor treatment, or termination of treatment for other reasons specified in the protocol. The maximum treatment duration for cadonilimab is 6 months.
  Interventions: Drug: Cadonilimab (AK104)

INTERVENTIONS:
Drug: Cadonilimab (AK104) — Patients with hepatocellular carcinoma after curative hepatectomy would receive cadonilimab 10 mg/kg intravenous infusion (dissolved in 0.9% NaCl 250 mL, within 60 minutes) Q3W, until disease progression, death, intolerance to toxicity, withdrawal of informed consent, initiation of new anti-tumor treatment, or termination of treatment for other reasons specified in the protocol. The maximum treatment duration for cadonilimab is 6 months.

SUMMARY:
This study aims to compare the safety and tolerability of cadonilimab applied after curative hepatectomy for hepatocellular carcinoma combined with high - risk recurrent factors.

DETAILED DESCRIPTION:
Hepatectomy and local ablation are the main curative treatment methods for hepatocellular carcinoma, but the 5-year recurrence rate after surgery is as high as 70%, which is the main bottleneck problem affecting the long-term prognosis of patients. This study aims to investigate the safety and tolerability of cadonilimab (PD-1/cytotoxic T lymphocyte antigen-4 (CTLA-4) bispecific antibody) applied after curative hepatectomy for hepatocellular carcinoma combined with high - risk recurrence factors.

ELIGIBILITY:
Inclusion Criteria:

* Sign a written informed consent before the implementation of any trial-related procedures.
* Male or female, aged ≥18 years and ≤70 years.
* ECOG PS score is 0 - 1 point.
* Subjects diagnosed with hepatocellular carcinoma by imaging criteria and/or pathology and who have received curative resection.
* The definition of curative resection complies with the definition of curativeness in the 2024 edition of the Chinese Guidelines for Primary Liver Cancer (CNLC).
* The postoperative recurrence risk stratification conforms to the high - risk group in the ERASL - pre or ERASL - post formula.
* No prior systemic antitumor treatment for hepatocellular carcinoma has been received.
* Child - Pugh liver function score of grade A or B7.
* Expected survival time > 6 months.

Exclusion Criteria:

* Previously diagnosed by histology/cytology, including fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, etc.
* Subjects with other malignant tumors within 5 years before enrollment, except for HCC. Subjects with other malignant tumors that have been cured by local treatment are not excluded, such as basal or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix or breast.
* History of hepatic encephalopathy or liver transplantation.
* Portal vein trunk or mesenteric superior vein, inferior vena cava tumor thrombus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 2 years
  the recurrence-free survival would be calculated and compared among different groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangxi Medical University Cancer Hospital, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Further enquiries can be directed to the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the full apper is publicated.

REFERENCES:
- [Background] Yuan G, Chen Y, Zhu P, Deng Q, Su K, Liu J, Wang Y, Li R, Li W, Zang M, Hu X, Wang JJ, Li Q, Du Y, Chen J. Cadonilimab (PD-1/CTLA-4) in combination with lenvatinib in unresectable hepatocellular carcinoma (uHCC): A retrospective real-world study. Heliyon. 2024 Sep 16;10(19):e37616. doi: 10.1016/j.heliyon.2024.e37616. eCollection 2024 Oct 15. PMID 39398001
- [Background] Wu X, Sun Y, Yang H, Wang J, Lou H, Li D, Wang K, Zhang H, Wu T, Li Y, Wang C, Li G, Wang Y, Li D, Tang Y, Pan M, Cai H, Wang W, Yang B, Qian H, Tian Q, Yao D, Cheng Y, Wei B, Li X, Wang T, Hao M, Wang X, Wang T, Ran J, Zhu H, Zhu L, Liu X, Li Y, Chen L, Li Q, Yan X, Wang F, Cai H, Zhang Y, Liang Z, Liu F, Huang Y, Xia B, Qu P, Zhu G, Chen Y, Song K, Sun M, Chen Z, Zhou Q, Hu L, Abulizi G, Guo H, Liao S, Ye Y, Yan P, Tang Q, Sun G, Liu T, Lu D, Hu M, Wang ZM, Li B, Xia M. Cadonilimab plus platinum-based chemotherapy with or without bevacizumab as first-line treatment for persistent, recurrent, or metastatic cervical cancer (COMPASSION-16): a randomised, double-blind, placebo-controlled phase 3 trial in China. Lancet. 2024 Oct 26;404(10463):1668-1676. doi: 10.1016/S0140-6736(24)02135-4. Epub 2024 Oct 16. PMID 39426385